CLINICAL TRIAL: NCT03731208
Title: Future Patient - Telerehabilitation of Patients After Knee Surgery
Brief Title: Telerehabilitation of Patients After Knee Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Mohammad Reza Naeemabadi, Principal Investigator, Laboratory for Welfare Technologies - Telehealth & Telerehabilitation, Integrative Neuroscience Research Group, SMI, Department of Health Science and Technology, Faculty of Medicine, Aalborg University, Aalborg, Denmark, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N-20180012
Record Dates: First submitted 2018-09-22; First posted 2018-11-06 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Knee Osteoarthritis
Keywords: Quality of life; Telerehabilitation; Knee rehabilitation; Knee Osteoarthritis; Total Knee Replacement
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): The patient assign to this arm receive the telerehabilitation program for 8-week after a knee operation
  Interventions: Device: Telerehabilitation

INTERVENTIONS:
Device: Telerehabilitation — The telerehabilitation program equipment consists of the following devices:
  * a tablet with a keyboard and a fingerprint sensor
  * two wearable sensors
  * a wireless modem
  * measuring tape

SUMMARY:
This project is aimed to investigate the feasibility of employing communication and sensor technologies for the patient after a knee operation.

In the study, it is hypothesized that the effectiveness of postoperative rehabilitation programs might be improved by establishing electronic communication between healthcare professionals and the patients. It is also believed that users satisfaction and patients quality of life will be improved.

The telerehabilitation program promises a synchronized communication as well as an individualized training program (by health professionals) based on the patient's electronic reports.

DETAILED DESCRIPTION:
Aim The objectives of this project are to assess the feasibility of using a telerehabilitation program for patients after a knee operation and investigate the acceptance of the provided solution by the patients and healthcare professionals.

Hypothesis It is hypothesized that the acceptance and satisfaction of patients and healthcare professionals by using the telerehabilitation program will be high and correlated with patients' exercise adherence and health recovery.

Telerehabilitation Group (Target Group) The subjects will be recruited before the operation and will be followed during an 8-week rehabilitation period.

In addition to the telerehabilitation program, the subjects will receive the regular treatment offered by Farsø Hospital in connection with total knee replacement surgery and are to follow the same rehabilitation procedure as regular patients (see below).

Before the operation, the project physiotherapist will hand over the telerehabilitation system equipment and instruct the subject how to use the system. In addition, the physiotherapist will also ask the subject to follow the instruction process and try the available services a few times. The physiotherapist makes sure that the subject can operate the system easily and without any challenges.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18
* Successful primary total knee replacement surgery at Farsø Hospital
* Referred to the regular rehabilitation program (self-training at home) by the physiotherapists at Farsø Hospital
* Ability to walk (with or without walking aids)
* Able to use electronic technologies and devices (for example: smart phone, tablet) or at least one relative who can assist in this matter
* Living in The North Denmark Region

Exclusion Criteria:

* Previous or current drug addiction defined as the use of cannabis, opioids or other drugs
* Previous or current neurologic, musculoskeletal or mental illnesses
* Any other aggravating medical complication (such as infection or DVT)
* Lack of ability to understand and accept trial procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Usability of the telerehabilitation program: semi-structured interview | The interview is conducted two weeks after discharge.
  The data is collected by a semi-structured interview
Exercise adherence | Everyday, started after discharge and for period of 8-weeks
  Measured by telerehabilitation system reports

SECONDARY OUTCOMES:
Self-reported pain, stiffness, and physical function: KOOS | After discharge (weeks 2, 8)
  Measured using Knee injury and Osteoarthritis Outcome Score (KOOS)
Self-reported pain and physical function: OKS | Baseline (before operation), and after discharge (weeks 0,2,4,6,8)
  measured by an electronic version of Oxford Knee Score (OKS)
Self-reported pain: VAS | Baseline (before operation), and every third day after discharge (for period of 8 weeks)
  Measured by an electronic report of the visual analog scale (VAS) of pain [minimum 0, Maximum 10] higher values represent a higher level of pain
Self-reported knee swelling | Baseline (before operation), and every third day after discharge (for period of 8 weeks)
  measured by an electronic report of knee circumference
Quality of life: EQ-5D | After discharge (weeks 2, 8)
  Measured using Euro Quality of Life - 5 Dimension (EQ-5D)
Users satisfaction: semi-structured interview | The interview is conducted two weeks after discharge.
  Measured by semi-structured interview

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Aalborg University, Aalborg
  - Aalborg University Hospital, Farsø

IPD SHARING:
Plan to Share IPD: No
No plan for sharing protocol was considered.